CLINICAL TRIAL: NCT02785432
Title: The Use of Low Level Laser Therapy With Physical Therapy for Pain and Improved Function in Individuals With Chronic Musculoskeletal Pain
Brief Title: Low Level Laser Therapy With Physical Therapy for Chronic Musculoskeletal Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty controlling for confounding factors
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ross Querry, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 012016-003
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham low level laser (Sham Comparator): Treatment will be administered 2x/w x 4 weeks as a standalone, then 2 times/week x 4 weeks in conjunction with standard physical therapy and counseling. The clinician will apply 10 minutes of low level laser therapy at a dosage of 0 watts for a total of 0 joules based on body surface area treated. Application will be with light to moderate contact pressure based on patient tolerance (should be no additional discomfort from laser). Area for administration will include 6 minutes of application along spine (C2-S1), and 4 minutes of application either to bilateral upper extremity or bilateral lower extremity based on areas of primary pain complaint. The contact head applicator will be used if soft tissue contact is tolerable. Otherwise, the non-contact head will be utilized.
  Interventions: Device: Sham low level laser
- Active low level laser (Active Comparator): Treatment will be administered 2x/w x 4 weeks as a standalone, then 2 times/week x 4 weeks in conjunction with standard physical therapy and counseling. The clinician will apply 10 minutes of low level laser therapy at a dosage of 15-25 watts for a total of 9,000-15,000 joules based on body surface area treated. This equates to standard acceptable dosing of 6-10 j/cm2 over the larger area of treatment. Application will be with light to moderate contact pressure based on patient tolerance (should be no additional discomfort from laser). Areas for administration and contact will otherwise be consistent with the sham group.
  Interventions: Device: Active low level laser

INTERVENTIONS:
Device: Sham low level laser — Sham laser will be administered using the same time and contact exposure as delivered for the active group, but without any energy delivered.
  Arms: Sham low level laser
Device: Active low level laser — Active treatment will be delivered using the time, contact, and energy exposures described in the arm description.
  Arms: Active low level laser

SUMMARY:
1. Examine the use of low level therapeutic laser (LLLT) combined with physical therapy for improvements in pain, range of motion, and function in individuals with chronic pain from musculoskeletal conditions.
2. Compare changes in pain, mobility, and ability to return to home/work/recreational activities between treatments with standard physical therapy plus LLLT or the standard physical therapy program alone.

DETAILED DESCRIPTION:
Potential subjects will be identified by their physician referral to the pain program and after initial evaluation by the medical personnel and physical therapy for appropriate inclusion in the pain program. For individuals who meet entry parameters for the pain program, this project will be discussed by their physical therapist for consideration of voluntary participation. If participants are willing to participate, appropriate consent and HIPPA permissions will be obtained.

After consent, the patient will be randomized to one of the two treatment cohorts which consists of utilizing either laser or sham laser before and during pain program participation. The principle investigator will be blinded to the treatment allocation group. The treating clinician will be aware of their treatment allocation assignment for laser application. Each treatment cohort will be completed as assigned. Physical therapy treatment in addition to the study intervention will be selected by the treating clinician based on participant's specific needs as standard of care would dictate. Outcome measures will be collected as described below.

Testing Schedule:

The assigned study intervention (LLLT or Sham) will be administered on each of the clinical visits for phase 1 and 2 of the study. Outcome measures will be completed on the following schedule.

Phase 1: Conducted during the period between acceptance to pain program and start the of the pain program (4 weeks). Baseline testing will be completed at the time of initial evaluation and enrollment to the study.

Phase 1 final testing (4 weeks) will be on the first clinic visit of the formal pain program. Phase 2: This phase is the 4-week formal pain program (2 visits/week x 4 weeks, total 8 visits). Final testing (8 weeks) will be on the final visit of the formal pain program.

Measurements:

A. Numerical pain rating scale (NPRS): perceived pain on scale of 0-10 (0=no pain, 10= extremely severe pain). Pain during the previous 24-hour period (best, worst, current) will be measured at baseline, 4 weeks, and 8 weeks. The average of 3 scores will be used.

B. Region specific functional outcome measure: A valid and reliable outcome tool of broad based physical function based on the body region of interest will be completed. Measured at baseline, 4 weeks, and 8 weeks.

C. Questionnaires of fear avoidance (FABQ, or TKS) and sleep quality (Pittsburg sleep index) will be taken as measures of quality of life and impact. Measures will be taken at baseline, 4 weeks, and 8 weeks.

All procedures, measurements, and interventions (exercises) are considered to be standard of care for rehabilitation and the subject's needs. The experimental aspect of the study is derived from the randomized selection of which laser intervention will be utilized before and during program participation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Primary referral and acceptance to the UTSW McDermott Multidisciplinary Pain Management Program. All diagnoses will be included.
3. Physical therapy specific inclusion for acceptance to the pain program (and this study) include:

   1. Musculoskeletal pain greater than 3 months
   2. Pain upon palpation or with movement of the extremities
   3. Medically cleared for physical therapy (exercise) in terms of cardiac, orthopedic, neurological impairments.
4. Cognitive, verbal, and physical abilities to self-detect and report pain and changes in exercise effort.
5. Ability to speak English and follow exercise based instructions.
6. Able to give informed consent.

Exclusion Criteria:

1. Inability to meet inclusion criteria for pain program
2. Current use of photosensitive medication (has been instructed to minimize sun exposure)
3. Active metastasis
4. Active infection
5. Diagnoses that exclude PT including cauda equine syndrome, myopathy, acute fracture (8-weeks).
6. Impaired sensation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Querry, PT, PhD, Principal Investigator — UT Southwestern
Locations (1):
- McDermott Pain Management Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Low Level Laser: Treatment will be administered 2x/w x 4 weeks as a standalone, then 2 times/week x 4 weeks in conjunction with standard physical therapy and counseling. The clinician will apply 10 minutes of low level laser therapy at a dosage of 15-25 watts for a total of 9,000-15,000 joules based on body surface area treated. This equates to standard acceptable dosing of 6-10 j/cm2 over the larger area of treatment. Areas for application and contact will otherwise be consistent with the sham group.
Period: Overall Study
Arm/Group | Sham Low Level Laser | Active Low Level Laser
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Low Level Laser | Active Low Level Laser | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (15.1) | 64.6 (15.8) | 60.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 11
Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Perceived pain on scale of 0-10 (0=no pain, 10= extremely severe pain).
  units on a scale | 4.0 (1.2) | 3.7 (0.96) | 3.9 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Perceived pain on scale of 0-10 (0=no pain, 10= extremely severe pain). Pain during the previous 24-hour period (best, worst, current) will be measured at T1-T8. The average of 3 scores will be used.
Time Frame: Baseline, 4 week, 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Low Level Laser | Active Low Level Laser
Number analyzed (Participants) | 4 | 7
score on a scale
  Baseline | 4 (1.2) | 3.7 (0.96)
  4 week | 6.1 (2.0) | 4.1 (1.2)
  8 week | 4.04 (1.4) | 3.6 (0.95)
Statistical Analysis 1: Comparison: Sham Low Level Laser vs Active Low Level Laser; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney) — Between group comparison at 8 weeks

2. Secondary Outcome: Tampa Scale of Kinesiophobia
Description: Valid and reliable 11 item assessment of kinesiophobia. Scores range from 11-44, with higher scores indicating greater degrees of kinesiophobia.
Time Frame: Baseline, 4 week, 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Low Level Laser | Active Low Level Laser
Number analyzed (Participants) | 4 | 7
score on a scale
  Baseline | 33 (1.1) | 27.5 (3.8)
  4 week | 31 (8.2) | 28.1 (6.5)
  8 week | 20.2 (9.2) | 22 (3.5)
Statistical Analysis 1: Comparison: Sham Low Level Laser vs Active Low Level Laser; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — Between group comparison at 8 weeks

3. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  The sum of scores for these seven components yields one global score. each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: Baseline, 4 week, 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Low Level Laser | Active Low Level Laser
Number analyzed (Participants) | 4 | 7
score on a scale
  Baseline | 9.75 (3.8) | 9.25 (5.2)
  4 week | 11.5 (6.1) | 9 (4.5)
  8 week | 9.75 (5.2) | 8 (4)
Statistical Analysis 1: Comparison: Sham Low Level Laser vs Active Low Level Laser; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney) — Between group comparison at 8 weeks

4. Secondary Outcome: Patient Specific Functional Scale
Description: Valid and reliable measure of the degree of difficulty with 3 self-selected activities as rated on an 11 point scale. The scores for the three activities are summed to create a total score ranging from 0-30, with higher scores indicating better/normal function.
Time Frame: Baseline, 4 week, 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Low Level Laser | Active Low Level Laser
Number analyzed (Participants) | 4 | 7
score on a scale
  Baseline | 11.5 (9.1) | 11.8 (3.5)
  4 week | 11.5 (9.1) | 9.7 (4.6)
  8 week | 13.8 (4.2) | 13.7 (5.2)
Statistical Analysis 1: Comparison: Sham Low Level Laser vs Active Low Level Laser; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney) — Between group comparison at 8 weeks

ADVERSE EVENTS:
Arm/Group | Sham Low Level Laser | Active Low Level Laser
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes